CLINICAL TRIAL: NCT05646589
Title: Implementation and Evaluation of a Person-centred Care Transition Support for People With Stroke/TIA
Brief Title: A Person-centred Care Transition Support for People With Stroke/TIA
Acronym: Missing Link
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Forte (Industry)
Responsible Party: Principal Investigator, Charlotte Ytterberg, Lecturer, associate professor (docent), Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022-02105-01
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: clinical trial; complex intervention; care transition; process evaluation; secondary prevention; hospital discharge; health literacy
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centred care transition support (Experimental): Person-centred dialogue intended to permeate all patient-provider communication, various pedagogical modes of information, a person-centred care and rehabilitation plan, and a bridging e-meeting to prepare patients for homecoming.
  Interventions: Behavioral: Person-centred care transition support
- Regular care transition (Active Comparator): Electronic referral from hospital healthcare professionals to the receiving neurorehabilitation team
  Interventions: Behavioral: Regular care transition

INTERVENTIONS:
Behavioral: Person-centred care transition support — Person-centred dialogue intended to permeate all patient-provider communication, various pedagogical modes of information, a person-centred care and rehabilitation plan, and a bridging e-meeting to prepare patients for homecoming.for persons who are to be discharged from hospitals after stroke or TIA
  Arms: Person-centred care transition support
Behavioral: Regular care transition — Regular care transitions, initiated by an electronic referral from hospital healthcare professionals to the receiving neurorehabilitation team
  Arms: Regular care transition

SUMMARY:
The goal of this clinical trial is to test a person-centred care transition support in people with stroke/TIA. The main questions it aims to answer are:

* Does a multi-component care transition intervention have an effect on perceived quality of care transitions, health literacy, collected medications, medication adherence, perceived person-centeredness, functioning, recurrent stroke/TIA, healthcare utilization and caregiver burden?
* What are the experiences of the intervention components and the implementation process?
* How does the intervention get adapted and implemented in practice?
* What contextual moderators and mechanisms of the intervention can likely explain the potential effects of the intervention?

Participants will receive a person-centred care transition support that includes a set of activities targeting how healthcare professionals can improve quality with care transition and support health literacy for self-management of secondary stroke prevention for persons who are to be discharged from hospitals after stroke or TIA.

Researchers will compare participants who receive the person-centred care transition support with participants receiving regular care transitions to see if the person-centred care transition support has any effects on perceived quality of care transitions, health literacy, collected medications, medication adherence, perceived person-centeredness, functioning, recurrent stroke/TIA, healthcare utilization and caregiver burden.

DETAILED DESCRIPTION:
Care transitions following a stroke call for integrated care approaches to reduce death and disability. The proposed research described in this study protocol aims to evaluate the ef-fectiveness of a person-centred multicomponent care transition support and the process in terms of contextual moderators, implementation aspects and mechanisms of impact.

A non-randomized controlled trial design will be used. The intervention includes person-centred dialogue intended to permeate all patient-provider communication, various pedagogical modes of information, a person-centred care and rehabilitation plan, and a bridging e-meeting to prepare patients for homecoming.

Patients with stroke or TIA who are to be discharged from the participating hospitals to home and referred to a neurorehabilitation team for continued rehabilitation will be included. Follow-ups will be conducted at one week, 3 months and 12 months. Data will be collected on the primary outcome of perceived quality of the care transition, and on the secondary outcomes of health literacy, medication adherence, and perceived person-centeredness. Data for process evaluation will be collected through semi-structured interviews, focus groups, partici-patory observations, and the Normalisation Measure Development Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients who have had a first time ever or recurrent stroke or TIA; who are to be discharged from the participating hospitals to home and referred to a neurorehabilitation team for continued rehabilitation; and who are able to give informed consent by themselves.

Exclusion Criteria:

* unable to give informed consent, due to e.g., severe aphasia or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Care Transition Measure | 1 week after discharge from hospital
  Questionnaire that assesses perceived quality in care transitions. The total score (0-100) reflects the overall perceived quality of the care transition, with lower scores indicating a poor quality care transition, and higher scores indicating a higher quality care transition

SECONDARY OUTCOMES:
The Medication Adherence Report Scale (patient) | 1 week, 3 and 12 months after inclusion
  Questionnaire that consists of 5 items that assesses medication adherence. Participants are asked to rate the frequency with which they engaged in each of the adherence-related behaviours on a five-point scale, where 5 = never, 4 = rarely, 3 = sometimes, 2 = often and 1 = always. Scores for each item were summed to give a total score, with higher scores indicating higher levels of reported adherence.
General Person-centred Care Questionnaire | 1 week, 3 and 12 months after inclusion
  Questionnaire with 21 questions about experiences of care and treatment. Responses are graded on a five-point Likert scale where a higher score represents a more person-centred experience i.e., a better outcome
Stroke Impact Scale, perceived recovery (patient) | inclusion, 1 week, 3 and 12 months after inclusion
  Perceived recovery after stroke is rated on a visual analogue scale ranging from 0 (no recovery) to 100 (full recovery)
Stroke Patient Education Retention | 1 week, 3 and 12 months after inclusion
  Questionnaire with five questions. scores range from 0 to 10 where a higher score represents a higher comprehension and retention of poststroke care education
EuroQol 5D | 1 week and 12 months after inclusion
  EuroQol 5D, consists of the EQ-5D Index and the EQ Visual Analog Scale. The EuroQol 5D comprises 5 pre-defined dimensions: Mobility, Self-care, Usual activities, Pain/discomfort and Anxiety/depression. The respondent rates each dimension on a three level scale as having no problem, a moderate problem or a severe problem. The answers are then converted to an index value (the EQ Index) ranging from 0 (representing death) to 1 (full health). The EQ VAS records the respondent's self-rated health on a 20-centimeter vertical visual analog scale with end-points ranging from 0 to 100. The single global question in the EQ VAS asks the individual to label his/her health as "the worst health you can imagine" (0) to "the best health you can imagine"
Health Literacy Survey | 1 week, 3 and 12 months after inclusion
  Questionnaire comprising 16 items focusing on four dimensions: ability to access/obtain health information, understand health information, ability to process/appraise health information, and ability to apply/use health information. Score ranges from 0-16 where a higher score represents a higher health literacy
Satisfaction with care and rehabilitation | 1 week, 3 and 12 months after inclusion
  Questionnaire with two questions. The respondent is asked to disagree or disagree with two statements on a Likert scale from 1 to 5 where a higher score represents higher satisfaction with care and rehabilitation
General Self-Efficacy Scale | 12 months after inclusion
  Questionnaire that assesses the strength of an individual's belief in his/her own ability to respond to novel or difficult situations and to deal with any associated obstacles or setbacks. The scale consists of 10 items rated on a four-point Likert scale ("not at all true" to "exactly true"). Means are calculated as the sum of all answers divided by ten (i.e., the total number of items)
Caregiver Burden Scale (significant other) | 3 months after inclusion
  Questionnaire that consists of 22 items for different types of subjective caregiver burden, covering areas of the caregiver's health, feelings of psychological well-being, relations, social network, physical workload, and environmental aspects. The items are scored on a scale from 1 to 4 and the higher the score the greater the burden.
Life Satisfaction Checklist, item 1 (significant other) | 3 months after inclusion
  Questionnaire that assesses life satisfaction with one global item "Life as a whole". Answering alternatives range from 1 (very dissatisfied) to 6 (very satisfied)
EuroQol 5D (significant other) | 3 months after inclusion
  Questionnaire consisting of the EQ-5D Index and the EQ Visual Analogue Scale. The EuroQol 5D-5L comprises five pre-defined dimensions: Mobility, Self-care, Usual activities, Pain/discomfort and Anxiety/depression. The respondent rates each dimension on a five level scale as having no problem, slight problems, moderate problem, severe problem, unable or extreme. The answers are then converted to an index value (the EQ Index) ranging from 0 (representing death) to 1 (full health). The EQ VAS records the respondent's self-rated health on a 20-centimeter vertical visual analo,g scale with end-points ranging from 0 to 100. The single global question in the EQ VAS asks the individual to label his/her health as "the worst health you can imagine" (0) to "the best health you can imagine"
Health Literacy Questionnaire | 1 week, 3 and 12 months after inclusion
  Questionnaire that assesses health literacy. The Health Literacy Questionnaire contains 44 items, which are divided into nine areas of health literacy. The first five scales are scored on a 4-point Likert scale (ranging from strongly disagree to disagree, agree, and strongly agree), building part I. The other four scales, representing part II, are scored on a 5-point Likert scale where respondents are asked to rate the level of difficulty in undertaking a task (ranging from cannot do, always difficult, usually difficult, sometime difficult, usually easy, and always easy). Higher scores indicate better health literacy.

OTHER OUTCOMES:
Patient Health Questionnaire-2 | inclusion, 1 week, 3 and 12 months after inclusion
  Questionnaire with to items that inquire about the frequency of depressed mood and anhedonia over the past two weeks. Score ranges from 0 (not at all) to 6 (nearly every day)
Fatigue visual analogue scale | inclusion, 1 week, 3 and 12 months after inclusion
  A visual analogue scale ranging from 0 (no fatigue) to 100 (extreme fatigue)
Barthel Index | inclusion, 1 week, 3 and 12 months after inclusion
  Questionnaire that includes 10 personal care and mobility activities, each scoring 0, 5 or 10 points resulting in a total score of 0 to 100, where a higher score reflects a greater degree of independence.
Modified Rankin Scale | 1 week, 3 and 12 months after inclusion
  Assesses degree of disability. Scores range from 0 (no disability) to 6 (death)
Montreal Cognitive Assessment Scale | inclusion, 3 and 12 months after inclusion
  Questionnaire assessing cognitive function. The scores range from 1 to 15 where 15 represents no cognitive impairment

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Aleris Dalengeriatriken, Stockholm
  - Danderyd hospital, Stockholm
  - Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results in a publication, after deidentification.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Immediately following publication and ending two years after publication.
Access Criteria: Since data can indirectly be traced back to the study participants, according to the Swedish and EU personal data sharing legislation, access can only be granted upon request. Request for access to the data can be put to our Research Data Office (rdo@ki.se) at Karolinska Institutet, and will be handled according to the relevant legislation. In most cases, this will require a data processing agreement or similar with the recipient of the data.

REFERENCES:
- [Background] Flink M, Lindblom S, Tistad M, Laska AC, Bertilsson BC, Warlinge C, Hasselstrom J, Elf M, von Koch L, Ytterberg C. Person-centred care transitions for people with stroke: study protocol for a feasibility evaluation of codesigned care transition support. BMJ Open. 2021 Dec 23;11(12):e047329. doi: 10.1136/bmjopen-2020-047329. PMID 34949604
- [Background] Hess Engstrom A, Flink M, Lindblom S, von Koch L, Ytterberg C. Association between general self-efficacy and health literacy among stroke survivors 1-year post-discharge: a cross-sectional study. Sci Rep. 2024 Mar 27;14(1):7308. doi: 10.1038/s41598-024-57738-z. PMID 38538651
- [Result] Flink M, Lindblom S, von Koch L, Carlsson AC, Ytterberg C. Health literacy is associated with less depression symptoms, higher perceived recovery, higher perceived participation, and walking ability one year after stroke - a cross-sectional study. Top Stroke Rehabil. 2023 Dec;30(8):865-871. doi: 10.1080/10749357.2023.2178133. Epub 2023 Feb 21. PMID 36803670
- [Result] Lindblom S, Ytterberg C, Flink M, Carlsson AC, Stenberg U, Tistad M, von Koch L, Laska AC. The Use of Teach Back at Hospital Discharge to Support Self-Management of Prescribed Medication for Secondary Prevention after Stroke-Findings from A Feasibility Study. Healthcare (Basel). 2023 Jan 30;11(3):391. doi: 10.3390/healthcare11030391. PMID 36766966
- [Result] Lindblom S, Tistad M, Flink M, Laska AC, von Koch L, Ytterberg C. Referral-based transition to subsequent rehabilitation at home after stroke: one-year outcomes and use of healthcare services. BMC Health Serv Res. 2022 May 3;22(1):594. doi: 10.1186/s12913-022-08000-7. PMID 35505404
- [Result] Lindblom S, Flink M, Elf M, Laska AC, von Koch L, Ytterberg C. The manifestation of participation within a co-design process involving patients, significant others and health-care professionals. Health Expect. 2021 Jun;24(3):905-916. doi: 10.1111/hex.13233. Epub 2021 Mar 17. PMID 33729653
- [Result] Lindblom S, Flink M, Sjostrand C, Laska AC, von Koch L, Ytterberg C. Perceived Quality of Care Transitions between Hospital and the Home in People with Stroke. J Am Med Dir Assoc. 2020 Dec;21(12):1885-1892. doi: 10.1016/j.jamda.2020.06.042. Epub 2020 Jul 29. PMID 32739283
- [Result] Lindblom S, Ytterberg C, Elf M, Flink M. Perceptive Dialogue for Linking Stakeholders and Units During Care Transitions - A Qualitative Study of People with Stroke, Significant Others and Healthcare Professionals in Sweden. Int J Integr Care. 2020 Mar 25;20(1):11. doi: 10.5334/ijic.4689. PMID 32256255
- [Result] Hess Engstrom A, Lindblom S, Flink M, Soderberg S, von Koch L, Ytterberg C. Stroke survivors' health literacy is not associated with caregiver burden: a cross-sectional study. Sci Rep. 2025 Feb 8;15(1):4720. doi: 10.1038/s41598-025-89523-x. PMID 39922929
- [Result] Lindblom S, Flink M, von Koch L, Laska AC, Ytterberg C. Feasibility, Fidelity and Acceptability of a Person-Centred Care Transition Support Intervention for Stroke Survivors: A Non-Randomised Controlled Study. Health Expect. 2024 Oct;27(5):e70057. doi: 10.1111/hex.70057. PMID 39373138
- [Derived] Lindblom S, Flink M, von Koch L, Tistad M, Stenberg U, Elf M, Carlsson AC, Laska AC, Ytterberg C. A person-centred care transition support for people with stroke/TIA: A study protocol for effect and process evaluation using a non-randomised controlled design. PLoS One. 2024 Mar 14;19(3):e0299800. doi: 10.1371/journal.pone.0299800. eCollection 2024. PMID 38483869